CLINICAL TRIAL: NCT01588288
Title: Diagnosis Interest of Galectin 3 Dosage in Nodular and Multinodular Goiter Pretreatment
Brief Title: Galectin 3 Dosage in Diagnosis of Nodular and Multinodular Goiter
Acronym: Galectins
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2011/042/HP; 2011-A00569-32 (Registry Identifier: RCB)
Record Dates: First submitted 2012-04-25; First posted 2012-04-30 (Estimated); Last update posted 2016-10-10 (Estimated); Status verified 2016-10

CONDITIONS: Goiter, Nodular
Keywords: Diagnosis; Galectin 3; Puncture; Goiter, nodular; Surgery
MeSH Terms: conditions — Goiter, Nodular; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Galectin 3 dosage (Experimental): Preoperative Galectin 3 dosage in plasma and water rinse of the needle aspiration biopsy
  Interventions: Procedure: Galectin 3 dosage

INTERVENTIONS:
Procedure: Galectin 3 dosage — Preoperative Galectin 3 dosage in plasma and water rinse of the needle aspiration biopsy.

SUMMARY:
The investigators will dose galectin 3 in plasma and water rinse of the needle aspiration biopsy in patients with thyroid nodules. The investigators aim to show that preoperative dosage of the galectin 3 could provide good diagnosis of malignant versus benign thyroid cancer.

DETAILED DESCRIPTION:
Endogenous cell-surface galectins have recently gained interest as antigenic determinants of varied tumor tissue. They are also used as potential targets for antitumor therapy by coupling cytotoxic molecules or radioisotopes either with carbohydrate residues, or with antibodies antigalectines.

In addition, the plasma level dosage of galectin 3 seems possible and provides a diagnostic help in thyroid lesions and in monitoring squamous cell head and neck.

In a study on thyroid tumors, the sensitivity [Se] and specificity [Sp] of the plasma level was poor (just over 70%), but this study was conducted with a low and heterogeneous recruitment (70 patients). The inclusion of a greater number of patients with a better selection would better inform us about qualities of these diagnostic assays.

An additional argument would be the dosage of galectins in the water rinse of the needle aspiration biopsy. This study has never been made so far and there is no evidence to predict its sensitivity and specificity. The advantage is that galectin will not be "diluted" as would be the case in an assay done in the blood. Moreover, it would select candidates for dosage nodules, ie those whose size would impose, if it was a cancer, to resort to surgical treatment more extensive than originally planned. Indeed, compared to preoperative already existing metering "interesting" dosage would diagnose:

* with a good reliability (Se and Sp > 80%)
* a cancer requiring additional treatment (i.e. surgical revision to achieve a total thyroidectomy, accompanied by lymph node dissection) resulting in a higher risk of morbidity if reoperation.

The investigators therefore believe that preoperative galectin 3 dosage in plasma or in the puncture water rinse could have strong arguments pointing to a neoplastic to a full initial gesture in a single surgical step, a gesture much less risky and expensive.

In this study, patients benefit from routine monitoring of thyroid nodules according to current recommendations. For surgical patients only, the information about the intervention will be collected to know the final histological diagnosis.

Galectin 3 will be measured preoperatively in :

* plasma
* water rinse of FNA.

The diagnostic characteristics of the assays, sensitivity and specificity will be established relative to the reference method which is the histological analysis of the specimen (report) asserting the existence of a vesicular lineage tumor, benign (adenoma) or malignant (papillary or follicular).

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* 18 years old or more
* Patient with one or more thyroid nodules with the following definition :

A nodule is a circumscribed intraparenchymal expansive development. This is thus a structure that appears on two cuts perpendicular ovoid. a nodule is visible on ultrasound by their mass effect (contour deformation), its ultrasound contrast relative to adjacent parenchyma or by repression of vascular structures at its periphery (halo and cantilever)

* Indication for a cytopuncture, in the opinion of the investigator
* Definitive postoperative histological analysis confirming a benign or malignant tumor of vesicular lineage cells.
* Patient affiliated to the french public welfare system
* Patient who signed an informed consent

Exclusion Criteria:

* Simple goiter
* Thyroid dysfunction
* Hashimoto's thyroiditis
* Basedow's disease
* No surgery at the end of the study
* After definitive postoperative histological analysis : lymphoma, medullary thyroid carcinoma, anaplastic thyroid cancer, or focal Hashimoto's thyroiditis
* Pregnancy
* Major under guardianship,
* Person deprived from him administrative and judicial liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2012-09; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Sensitivity (Se) and specificity (Sp) of plasmatic galectin 3 dosage in preoperative | 1 day
  Se and Sp of plasmatic galectin 3 dosage will be established relative to the reference method which is the histological analysis of the specimen (report) asserting the existence of a vesicular lineage tumor, benign (adenoma) or malignant (papillary or follicular).
  The threshold giving the best compromise for the values of Se and Sp will be searched graphically. Then the area under the curve and its confidence interval at 95% will be calculated and will be tested against the value 0.5, that is to say an area where the assay has no diagnostic value.

SECONDARY OUTCOMES:
Sensitivity (Se) and specificity (Sp) of preoperative galectin 3 dosage in the water rinse of the needle aspiration biopsy | Once in preoperative
  Se and Sp of galectin 3 dosage in the water rinse of the needle aspiration biopsy will be established relative to the reference method which is the histological analysis of the specimen (report) asserting the existence of a vesicular lineage tumor, benign (adenoma) or malignant (papillary or follicular).
  The threshold giving the best compromise for the values of Se and Sp will be searched graphically. Then the area under the curve and its confidence interval at 95% will be calculated and will be tested against the value 0.5, that is to say an area where the assay has no diagnostic value.

CONTACTS AND LOCATIONS:
Overall Officials: Anne CAILLEUX, MD, Principal Investigator — University Hospital, Rouen
Locations (2):
- France (2):
  - Centre Henri Becquerel, Rouen
  - CHRouen, Rouen